CLINICAL TRIAL: NCT02095080
Title: Determination of the Tolerable Upper Intake Level (UL) of Leucine in Healthy Elderly Men (70-75 Yrs)
Brief Title: Determination of the UL of Leucine in Healthy Elderly Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: International Council on Amino Acid Science (Other)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H14-00235
Record Dates: First submitted 2014-03-19; First posted 2014-03-24 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Elderly Men
Keywords: Leucine; Upper Intake Level (UL); Elderly; Amino acids; Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Leucine intake (Experimental): Dietary supplement: Leucine intake
  Interventions: Dietary Supplement: Leucine intake

INTERVENTIONS:
Dietary Supplement: Leucine intake — Oral consumption of eight hourly experimental meals- Includes 4 tracer-free experimental meals containing a mixture of free amino acids, calories from a flavored liquid and protein free cookies and 4- labeled amino acid experimental meals.

SUMMARY:
Amino acid are the building blocks of the body's protein. Some amino acids, including leucine, cannot be made in the body and must be obtained from diet, these are called essential. With increase in age the body's muscle mass decrease and studies have suggested that dietary supplementation of leucine may have potential health benefits in elderly in regards to prevention of age related loss of lean muscle mass, and thus may help improve the quality of life in elderly.

Currently, a safe upper dietary intake level of leucine has not been established for healthy elderly. Prior to exploring whether leucine supplementation will prevent or decrease loss of lean muscle mass in elderly we propose to identify the upper intake of leucine in healthy elderly.

The purpose of this study is to determine the tolerable upper intake level (UL) of leucine in healthy elderly men (70 - 75 yrs)

The investigators hypothesize that with a careful graded stepwise increase in leucine intake in elderly men, above the Estimated Average Requirement (EAR - 50 mg/kg/d), the body's ability to oxidize/dispose of excess amino acids will reach a maximum. With increased leucine intakes we hypothesize an increase in plasma ammonia concentrations and increases in plasma leucine and urinary leucine excretion.

ELIGIBILITY:
Inclusion Criteria:

* Men 70 - 75 years of age
* Free of chronic diseases including; sarcopenia, heart disease, kidney disorders, liver disease, chronic high blood pressure and or diabetes.
* Free of any cognitive disorders
* Men not enrolled in any other research studies
* Men who are not claustrophobic

Exclusion Criteria:

* Men not within the age 70 -75 years
* Men diagnosed with a chronic diseases including; sarcopenia, heart disease, kidney disorders, liver disease, chronic high blood pressure and/or diabetes
* Men allergic to milk, eggs and egg protein
* Men who are claustrophobic
* Men who are currently enrolled in other research studies

Ages: 70 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
13 carbon dioxide production | 8 hours (1 study day)
  Urine, plasma and breath samples will be collected during the study to measure the rate of oxidation of the tracer.

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, PhD, Principal Investigator — Child & Family Research Institute/University of British Columbia
Locations (1):
- Child & Family Research Institute, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Rasmussen B, Gilbert E, Turki A, Madden K, Elango R. Determination of the safety of leucine supplementation in healthy elderly men. Amino Acids. 2016 Jul;48(7):1707-16. doi: 10.1007/s00726-016-2241-0. Epub 2016 Apr 30. PMID 27138628